CLINICAL TRIAL: NCT04795661
Title: Immunotherapy in MSI/dMMR Tumors in Perioperative Setting.
Acronym: IMHOTEP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMHOTEP (ET20-093)
Record Dates: First submitted 2021-03-11; First posted 2021-03-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Localized Resectable Tumor; MSI/dMMR
Keywords: Oncology; MSI/dMMR status; Pembrolizumab; Immunotherapy; Phase II; Neoadjuvant treatment
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort Colorectal cancer (CRC) (Experimental): Pembrolizumab prior to surgery
  Interventions: Drug: Pembrolizumab
- Cohort Oesogastric cancer (Experimental): Pembrolizumab prior to surgery
  Interventions: Drug: Pembrolizumab
- Cohort Other cancer (Experimental): Pembrolizumab prior to surgery
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Administered intravenous (IV)
  Other Names: MK3475 - Keytruda®

SUMMARY:
This trial is a multicenter, 3-cohort, prospective, Phase II trial conducted in patients with untreated resectable MSI/dMMR carcinomas and aiming to evaluate the safety and the efficacy of ICI (immune checkpoint inhibitor) as neoadjuvant treatment in these patients.

We hypothesize that immune checkpoint inhibitors (ICPi) will benefit to MSI/dMMR tumors from the early stages, whatever their anatomical origin. We assume that this neoadjuvant treatment would improve the response rate, providing even high rate of pathological complete responses and prolong patients survival.

We anticipated colorectal and gastric cancers to be the most frequent recruited and constructed our statistical hypothesis with results in those 2 cancers. However patients with other localized MSI/dMMR tumors could be included.

DETAILED DESCRIPTION:
TREATMENT PLAN:

Pre-operative pembrolizumab will be administered intravenously (IV) over 30 minutes at the dose of 400 mg according to recent summary of product characteristics (SPC). Until four doses will be administered 6 weeks before the planned surgery, as close as possible to inclusion, and whenever possible during standard visit (surgery, anesthesia or other).

Surgery will be performed during the 6th week after the last pembrolizumab injection, as per standard practices.

An adjuvant treatment will be administered upon the Investigator decision, depending on the protocol: the results and tolerance of pre-operative treatment and ability of the patient to receive the treatment regarding his general post-operative condition.

STATISTICAL ANALYSIS:

A total of 240 patients will be enrolled in this study

Sample size was thus evaluated by analogy with an A'Hern's single stage phase II design with P0=25%, P1=50% and 85% power.

A sequential Bayesian design will be used to allow continuous monitoring of the primary endpoint and update knowledge gradually.

For each cohort, interim analyses are planned after 6-week follow up of the first 10 patients (i.e. after surgery) and then every 10 patients.

Early stopping will be recommended if there is a high posterior probability (≥90%) given observed data that the rate of pathological response is lower than 50%.

DATA ENTRY, DATA MANAGEMENT AND STUDY MONITORING:

All the data concerning the patients will be recorded in the electronic case report form (eCRF) throughout the study. Serious adverse event (SAE) and Adverse Event of Specific Interest (AESI) reporting will be also paper-based by e-mail and/or Fax.

The sponsor will perform the study monitoring and will help the investigators to conduct the study in compliance with the clinical trial protocol, Good Clinical Practices (GCP) and local law requirements.

ELIGIBILITY:
Inclusion criteria

I1. Age ≥ 18 years on the day of signing informed consent.

I2. Histologically proven localized non-metastatic tumor included in one of the 4 cohorts:

* Colon or rectal Cancer (cT3/T4 N0 M0 ou cT N+ M0) OR
* Oesogastric (gastric, gastro-oesophageal or oesophageal) cancer (cT2 to cT4 N M0) OR
* Other tumor types (cT2 to cT4 N M0): small bowel adenocarcinoma (duodenum, jejunum, ileum).

I3. MSI/dMMR established by immunohistochemistry (IHC) [MMR protein expression] and polymerase chain reaction (PCR) (or Next-Generation Sequencing (NGS)) [both techniques are required] and validated by coordinator's team.

MMR and/or MSI tumors will be assessed using IHC with four antibodies (anti-MLH1, anti-MSH2, anti-MSH6 and anti-PMS2) and PCR (pentaplex panel is recommended: BAT-25, BAT-26, NR-21, NR-24, and NR-27) prior to screening. Loss of MLH1 and PMS2 / or MSH2 and MSH6 / or MSH6 alone / or PMS2 alone protein staining by IHC indicates dMMR, and tumor with ≥ 2 unstable markers analyzed on PCR proves MSI/dMMR, NGS will be accepted instead of PCR analysis.

I4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 to 1 within 7 days prior to the inclusion.

I5. Adequate bone-marrow, hepatic, and renal functions, within 10 days prior to the start of study treatment with:

* Hemoglobin ≥ 9 g/dl or ≥ 5.6 mmol/l, neutrophils ≥ 1.0 x 109/l, platelets ≥ 100 x 109/l,
* Creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 30 ml/min/1.73m² using either MDRD or CKD-EPI formula,
* AST and ALT ≤ 3 x ULN, total bilirubin ≤ 1.5 ULN (or direct bilirubin ≤ ULN for patients with total bilirubin >1.5 × ULN),
* International normalized ratio (INR) OR prothrombin time (PT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants.

I6. Covered by a medical/health insurance.

I7. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

I8. Patients of childbearing potential accepting to use effective contraceptive measures or abstain from heterosexual activity, for the course of the study through 4 months after the last dose of pembrolizumab MK-3475 adjuvant treatment or 6 months after adjuvant chemotherapy or being surgically sterile. Refer to Appendix 1 for approved methods of contraception.

I9. Signed and dated IRB/IE approved informed consent form.

Non-inclusion criteria

E1. MSS/pMMR tumors.

E2. Metastatic disease (stage IV).

E3. HIV positive with CD4 count under 400 cells/mm3

E4.Concurrent active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] positive and/or detectable HBV DNA) or Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection).

E5. Active systemic autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin) is not considered a form of systemic treatment and is allowed.

E6. Interstitial lung disease.

E7. Prior (non-infectious) pneumonitis requiring systemic corticosteroid therapy or current pneumonitis.

E8. History of severe hypersensitivity to another monoclonal antibody.

E9. Receiving immunosuppressive therapy or having received corticosteroids (in dosing exceeding 10 mg daily of prednisone equivalent) within the last 2 months before inclusion.

E10. Active infections.

E11. Radiotherapy within the 2 weeks before inclusion. Patients must have recovered from all radiation related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease. - Not applicable

E12. Live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.

E13. Known history of active TB (Bacillus Tuberculosis).

E14. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.

E15. Pregnant or breastfeeding woman or patient expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 4 months after the last dose of study treatment.

E16. Patient requiring tutorship or curatorship.

E17. Ongoing anti-cancer treatment for another cancer (to be discussed with the coordinator in case of hormone therapy).

E18. Prior history of other malignancies (except for HNPCC or Lynch syndrome-related cancers) unless the subjects has been free of the disease for at least 2 years.

E19. Patient hospitalized at the moment of inclusion and treatment initiation (palliative care unit, retirement home … are considered as hospitals).

E20. Recent hemorrhage (in the month before inclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Rate of complete pathological response (pCR) after surgery | 6 weeks after first injection
  A complete pathological response will be defined as 0% viable tumor cells.

SECONDARY OUTCOMES:
Safety of the perioperative treatment | 60 Months (over the whole study)
  Safety profile, determined using the National Cancer Institute - Common Terminology Criteria for Adverse Event (NCI-CTC AE) grading scale version 5. Adverse events will be described by their intensity and severity
Rate of surgical complications (post-operative morbidity) | 1 Month after sugery
  The rate of surgical complications (post-operative morbidity) will be assessed according to modified Clavien Dindo scoring
Rate of patients with the R0 resection | 60 Months
  Percentage of patients with the R0 resection
Major pathological response rate | 60 Months
  Percentage of patients with major pathological response (≤ 10% residual viable tumor)
Recurrence-free survival (RFS) | 60 Months
  RFS defined as the time from the date of first study treatment administration to the date of first documented recurrence
Overall response rate (ORR) at 4, 10, 16 and 21 weeks after the pembrolizumab initiation | 4, 10, 16, 21 weeks after first study treatment injection
  Percentage of patients with objective response at week 4, 10, 16 and 21 (complete or partial response) after neoadjuvant pembrolizumab, according to RECIST v1.1.
Rate of second cancer in the Lynch syndrom spectrum | 60 Months
  Percentage of patients with second cancer
The overall survival (OS) | From 60 months
  OS, defined from the date of first study treatment administration to the date of death due to any cause.
Progression-free survival (PFS) after recurrence | 60 months
  PFS, defined from the date of first documented recurrence to the date of documented progression.
Quality of life (QoL) | Baseline,cycle 2 and 4 before surgery and 5 months after the surgery
  QoL, assessed using the EORTC QLQ-C30
The prognostic value of lung immune prognostic index (LIPI) | 60 months
the progression free survival for patient without surgery | 60 months
  PFS, defined from the date of first documented recurrence to the date of documented progression.

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Amiens Picardie, Amiens
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Centre Georges-Francois Leclerc, Dijon
  - Hopital Huriez, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut du Cancer Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - APHP Hôpital Saint-Louis, Paris
  - Institut mutualiste Montsouris, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - APHP - Hôpital Saint-Antoine, Paris
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - CHU Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - CHU Saint Etienne, Saint-Etienne
  - Centre Paul Strauss, Strasbourg
  - Institut de cancérologie Strasbourg Europe, Strasbourg